CLINICAL TRIAL: NCT05036213
Title: The Effects of Oral Inorganic Nitrate Supplementation on Lower Limb Perfusion and Metabolism During Exercise in Patients With Peripheral Arterial Disease (PAD)
Brief Title: The Effects of Oral Inorganic Nitrate Supplementation on Lower Limb Perfusion During Exercise in Patients With PAD
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Jason Allen, Professor in kinesiology, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 21774
Record Dates: First submitted 2021-09-01; First posted 2021-09-05 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Peripheral Arterial Disease; Peripheral Vascular Diseases
Keywords: PAD; nitrate; nitric oxide
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled, cross-over design. This means that all subjects will complete both supplementation phases in a randomized order.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dietary nitrate (Active Comparator): The active treatment, beetroot juice (BEET IT, James White Drinks, Ipswich, UK), contains 6.2mmol of inorganic nitrate. Participants will continue supplementation until they complete all testing visits.
  Interventions: Drug: BEET IT - Concentrate Beet root juice
- concentrated beet root juice with depleted nitrate content (Placebo Comparator): The placebo treatment is also beetroot juice provide by the same company (BEET IT, James White Drinks, Ipswich, UK), but it does not contain any inorganic nitrate. Participants will continue supplementation until they complete all testing visits.
  Interventions: Drug: BEET IT - Concentrate Beet root juice (nitrate depleted)

INTERVENTIONS:
Drug: BEET IT - Concentrate Beet root juice — Each bottle contains 75ml of concentrated beetroot juice with approximately 6.2mmol of inorganic nitrate. The product is provided by BEET IT, James White Drinks, Ipswich, UK.
  Other Names: Dietary Nitrate supplementation (nitrate rich)
  Arms: Dietary nitrate
Drug: BEET IT - Concentrate Beet root juice (nitrate depleted) — Each bottle contains 75ml of concentrated beetroot juice with depleted nitrate, thus, no inorganic nitrate is found in thisbeverage. The product is also provided by BEET IT, James White Drinks, Ipswich, UK.
  Other Names: Dietary Nitrate supplementation (nitrate depleted)
  Arms: concentrated beet root juice with depleted nitrate content

SUMMARY:
Peripheral arterial disease (PAD) is a highly prevalent and costly condition. Intermittent claudication (IC), defined as ischemic leg pain that occurs with walking, results in functional impairment, reduced daily physical activity, and a lower quality of life. Although the mechanisms contributing to functional impairment are not fully delineated, current evidence suggests that the uncoupling of skeletal muscle cellular metabolism from tissue perfusion may be responsible for exercise intolerance. We have previously shown increases in plasma inorganic nitrite, via oral nitrate, produced clinically significant increases exercise performance in patients with PAD+IC.

The hypothesis of this proposal is in patients with PAD+IC, 3-6 days of oral dietary nitrate consumption (in the form of concentrated beetroot juice) will produce a greater tissue perfusion, oxygen delivery, and enhanced muscle metabolism in comparison to placebo. This will translate into an increase in physical performance in both muscle specific plantar flexion exercise and treadmill measures of pain free ambulation. In order to test this hypothesis, we will recruit 10 patients PAD+IC in a randomized, double-blind, placebo controlled, cross over design.

DETAILED DESCRIPTION:
Peripheral Arterial Disease (PAD) is characterised by blockages (occlusion or stenosis) in the large arteries of the lower limbs. It is estimated that worldwide prevalence of PAD has increased by 23.5% in the last decade and now affects 202 million people. PAD prevalence increases with age from 5% of 45-49-year-old up to 19% in those >70years old and smoking and diabetes are causative factors. PAD is vastly understudied in comparison to cardiac or cerebrovascular diseases. Intermittent claudication (IC) is the major clinical manifestation of PAD and occurs when arterial occlusive disease reduces blood flow to the peripheral vasculature during exercise. Among subjects with intermittent claudication from PAD, 1/3rd have pain during light activity at home and an additional 1/3rd have pain walking a short distance (one block). These patients suffer from a markedly impaired quality of life and a high perception of disability. Increased pain free ambulation is a primary goal of therapy for PAD as this is related to improved quality of life.

Although the ankle-brachial systolic blood pressure index (ABI) and limb blood flow testing are used to diagnose PAD, most research studies fail to show a relationship between these measures and functional capacity. Confounding the understanding of this disease is that surgical revascularization, which improves blood flow, does not normalize exercise performance and ambulation can be increased without changes in hemodynamics. Professor Allen (PI) has previously shown increases in peak hyperemic leg blood flow with exercise training but failed to find a relationship between these changes and increases in claudication onset time (COT) and peak walk time (PWT). Professors Allen and Annex (Chief UVa Health System - Cardiovascular Medicine) have also shown increases in gastrocnemius capillary density following exercise training and a correlation with VO2peak. This suggests, in the presence of conduit vessel stenosis, patients become more reliant on the microvasculature to distribute available blood and oxygen to working tissues more efficiently.

Nitric Oxide (NO) is produced by the vascular endothelium and plays an important role in vasodilation, flow regulation and platelet function. Disruptions in the production of NO have been implicated in the pathogenesis of vascular disease. It was originally believed that the bioactivity of NO was limited both temporally and spatially to the proximity of the vascular endothelium where it was produced. It is now clear that several protected NO-derived species may be transported through the vasculature to be released at critical areas of the circulation, where it can influence macro- and micro-vascular tone and possibly vasculopathy. Under normal conditions, this endocrine-like role is precisely controlled: whereby during normoxia NO is conserved but under hypoxic conditions NO is liberated and can initiate vasodilation. One potential therapeutic option involves the conversion of inorganic nitrate (NO3-) and nitrite (NO2-) anions into NO (and other bioactive species). This is an attractive approach, as it is biologically distinct from endothelial-NO synthase and can be achieved easily via oral administration. Inorganic NO3- is abundant in green leafy vegetables, beets, celery, lettuce, radishes and spinach.

We were the first group to demonstrate acute increases in plasma NO2- concentration (using beetroot juice containing 9mM NO3-), and increased walking performance in subjects with PAD+IC. COT increased by 18% (32sec) and PWT by 17% (65sec). This is a clinically meaningful and statistically significant increase for a disease state characterized by reduced physical function and quality of life. There were no changes in ABI or endothelial function suggesting no increase in endogenous vascular NO. The increases in performance were accompanied by a reduction in fractional oxygen extraction at the working tissues, measured by near infra-red spectroscopy (NIRS) suggesting increased perfusion to working tissues.

We have subsequently demonstrated that chronic dosing in combination with 36 sessions of exercise training (EX+BR) also generated significant increases in pain free ambulation (COT) and like-wise reductions in deoxyhemoglobin during exercise, when compared to an identical exercise regimen coupled with placebo.

Unfortunately, while Near Infrared Spectroscopy (NIRS) data during a physiological challenge is indicative, it is also relatively imprecise -NIRS measures only relative oxygenation/deoxygenation for the whole tissue-bed. A much more precise non-invasive approach has been developed by Professor Christopher Kramer (UVa Health System - Cardiovascular Medicine, Noninvasive Cardiovascular Imaging) and Professor Craig H. Meyer (Department of Biomedical Engineering) which utilizes Pulsed Arterial Spin Labelling (PASL) coupled with a cuff occlusion or plantar flexion exercise stress test developed by Professor Arthur Weltman (UVa - Department of Kinesiology). This allows for the creation of tissue perfusion maps and differentiation between specific gastrocnemius muscle compartments in a spatial and temporally resolved fashion. Additionally, we will employ Creatine Exchange Saturation transfer (CrCEST) to measure PCr recovery kinetics after exhaustive exercise or until subjects symptoms limit their exercise tolerance.

These techniques in combination will allow us to differentiate deficits in tissue perfusion and metabolism (mitochondrial function) for specific compartments of the gastrocnemius muscle before and after intervention. The sensitivity to detect changes following inorganic nitrate (BR) supplementation was previously demonstrated in healthy subjects during severe exhaustive exercise (which creates hypoxic conditions in the tissue bed analogous to those in patients with PAD+IC during mild exercise). The participants on BR showed an increase in exercise tolerance and a reduction in PCr depletion, suggesting changes in muscle metabolism/function. However, the effect of BR on the metabolic responses and tissue perfusion during exhaustive exercise in PAD patients has not been investigated to date.

The hypothesis of this proposal is in patients with PAD+IC, 3-6 days of oral dietary nitrate consumption (in the form of concentrated BR) will produce a greater tissue perfusion, oxygen delivery, and enhanced muscle metabolism in comparison to placebo (PL). This will translate into an increase in physical performance in both muscle specific planter flexion exercise and treadmill measures of pain free ambulation. In order to test this hypothesis, the following specific aims will recruit 24 PAD+IC patients in a randomized, double-blind, placebo controlled, cross over design.

Aim 1. To determine between treatment differences (BR v PL) in phosphocreatine recovery time constant (PCr) measured by Creatine chemical Exchange Saturation Transfer (CrCREST).

Aim 2. To determine between treatment differences (BR v PL) in peak exercise, maximal hyperemia in different lower limb compartments (anterior, lateral, gastrocnemius, soleus and deep compartments) by Pulsed Arterial Spin Labelling (PASL).

Aim 3. To determine relations in between treatment changes in walking performance COT and PWT and lower limb compartmental perfusion characteristics (Aim 2) and phosphocreatine recover kinetics (Aim 1).

ELIGIBILITY:
Inclusion Criteria:

* - History of stable intermittent claudication for 3 or more months, and an Ankle-brachial index test (ABI) <0.9 at rest.
* Symptomatic PAD (claudication or critical limb ischemia)

Exclusion Criteria:

* - Limb threatening ischemia, including rest pain and/or gangrene; impending limb loss or chronic osteomyelitis.
* Lower extremity vascular surgery, angioplasty or lumbar sympathectomy within 3 months of enrollment;
* severe peripheral neuropathy or any condition other than PAD that limits walking such as unstable angina;
* history of significant left main or three vessel coronary artery disease (>70% stenosis, unprotected by grafts) or recent myocardial infarction (6 weeks);
* chest pain during treadmill exercise which appears before the onset of claudication,
* chronic renal failure with an eGRF<30; Type 1diabetes mellitus, a BMI>40, and a HbA1c>8.5%. Refusal to give or inability to give informed consent. Pregnancy (Self-reported).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Phosphocreatine kinetics after maximal exercise | After a minimum of 3 days of supplementation with either Placebo or nitrate rich beverage.
  The primary outcomes to be analyzed will be treatment differences (BR v PL) in phosphocreatine recovery time constant (PCr) measured by Creatine chemical Exchange Saturation Transfer (CrCREST).
  The subjects will be positioned within the scanner feet first with the calf at the isocenter of the magnet and a flexible phased array coil will be positioned and wrapped around the calf of interest. Imaging of calf muscle energetics using creatine chemical exchange saturation transfer (CrCEST, no contrast agent used) will be performed after pedal ergometry until exhaustion or limiting symptoms

SECONDARY OUTCOMES:
Maximal hyperemia in different lower limb compartments | After a minimum of 3 days of supplementation with either Placebo or nitrate rich beverage.
  At the Prisma 3T scanner at Fontaine, subjects will be positioned within the scanner feet first with the calf at the isocenter of the magnet and a flexible phased array coil will be positioned and wrapped around the calf of interest. Subjects to complete plantar flexion ergometry to exhaustion or claudication. Imaging of calf muscle perfusion by arterial spin labeling (ASL, no contrast agent used) will be performed after pedal ergometry until exhaustion or limiting symptoms.
Peak exercise | After a minimum of 3 days of supplementation with either Placebo or nitrate rich beverage.
  Subjects will be tested on two different occasions (PL vs Beet root juice) for how long they can walk (in seconds) on a treadmill. The treadmill walking test is designed specifically for a claudication-limited population (i.e. the Gardner protocol). During this walking test the speed is maintain at 2mph with a 2%-grade increase every 2 minutes.
Claudication Onset Time | After a minimum of 3 days of supplementation with either Placebo or nitrate rich beverage.
  During the treadmill exercise protocol subjects will report when they start to feel pain in their lower limbs (or the affect leg).
Vascular Function - Brachial Flow Mediated Dilation | After a minimum of 3 days of supplementation with either Placebo or nitrate rich beverage.
  A high-resolution ultrasound will be used to capture images of the brachial artery at baseline, during 5 minutes of forearm occlusion, and for two minutes (with r-wave trigger) following occlusion cuff release. These data points will be utilized to calculate the percentage of change in brachial artery diameter following reactive hyperemia (occlusion release).
Vascular stiffness | After a minimum of 3 days of supplementation with either Placebo or nitrate rich beverage.
  Vascular stiffness will be assessed by measures of pulse wave velocity using applanation tonometry (SphygmoCor EXCEL system V1). The measures provided by PWA include: central systolic pressure (mmHg); central pulse pressure (PP) mmHg; augmentation pressure (AP) and augmentation index (AIx).
  Pulse wave velocity is measured via a simultaneous comparison of the carotid and femoral arterial pulses. A thigh cuff will be placed around the patient's upper thigh which acts to measure the femoral pulse via pulsations, whilst simultaneously a tonometer will be used to assess the carotid pulse. Higher pulse wave velocities from the carotid to femoral arteries indicates higher aortic stiffness.

CONTACTS AND LOCATIONS:
Overall Officials: Jason D. Allen, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this RCT, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 9 months and ending 36 months following article publication.

REFERENCES:
- [Background] Isbell DC, Epstein FH, Zhong X, DiMaria JM, Berr SS, Meyer CH, Rogers WJ, Harthun NL, Hagspiel KD, Weltman A, Kramer CM. Calf muscle perfusion at peak exercise in peripheral arterial disease: measurement by first-pass contrast-enhanced magnetic resonance imaging. J Magn Reson Imaging. 2007 May;25(5):1013-20. doi: 10.1002/jmri.20899. PMID 17410566
- [Background] Isbell DC, Berr SS, Toledano AY, Epstein FH, Meyer CH, Rogers WJ, Harthun NL, Hagspiel KD, Weltman A, Kramer CM. Delayed calf muscle phosphocreatine recovery after exercise identifies peripheral arterial disease. J Am Coll Cardiol. 2006 Jun 6;47(11):2289-95. doi: 10.1016/j.jacc.2005.12.069. Epub 2006 May 15. PMID 16750698
- [Background] Lopez D, Pollak AW, Meyer CH, Epstein FH, Zhao L, Pesch AJ, Jiji R, Kay JR, DiMaria JM, Christopher JM, Kramer CM. Arterial spin labeling perfusion cardiovascular magnetic resonance of the calf in peripheral arterial disease: cuff occlusion hyperemia vs exercise. J Cardiovasc Magn Reson. 2015 Feb 22;17(1):23. doi: 10.1186/s12968-015-0128-y. PMID 25890198
- [Background] Kenjale AA, Ham KL, Stabler T, Robbins JL, Johnson JL, Vanbruggen M, Privette G, Yim E, Kraus WE, Allen JD. Dietary nitrate supplementation enhances exercise performance in peripheral arterial disease. J Appl Physiol (1985). 2011 Jun;110(6):1582-91. doi: 10.1152/japplphysiol.00071.2011. Epub 2011 Mar 31. PMID 21454745